CLINICAL TRIAL: NCT04407845
Title: Etude de l'Incidence et Des Facteurs prédictifs de la Survenue de Fibrillation Atriale Sous Ibrutinib
Brief Title: Atrial Fibrillation in Patients Receiving Ibrutinib
Acronym: FABRIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: European Georges Pompidou Hospital (Other)
Responsible Party: Principal Investigator, Mariana Mirabel, MD, PhD, Associate Professor, European Georges Pompidou Hospital
Other Study IDs: 00011928 FABRIC
Record Dates: First submitted 2020-05-14; First posted 2020-05-29 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Leukemia, Chronic Lymphatic; Mantle Cell Lymphoma
Keywords: atrial fibrillation; haematology; systemic hypertension; prognosis; heart
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Atrial Fibrillation; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ibrutinib (a tyrosine kinase inhibitor targeting Bruton) is a standard of treatment in haematology. According to retrospective data, atrial fibrillation and systemic hypertension are common ibrutinib-related advserse events. The investigators aim at prospectively establishing the incidence of thesedrug related advsere events through clinical monitoring and attempt at identifying populations at risk.

ELIGIBILITY:
Inclusion Criteria:

* All patients deem to start ibrutinib therapy

Exclusion Criteria:

* Past history of ibrutinib therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective consecutive cohort
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-05-21 (Actual); Primary Completion 2022-05-21 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of cardiovascular events on ibrutinib | 6 months
  Evaluate the incidence of cardiotoxicity (composite endpoint) in a cohort of patients referred to a cardio-oncology before initiation of ibrutinib.

SECONDARY OUTCOMES:
Incidence of supra-ventricular arrythmias | 6 months
  Number of patients with supra-ventricular arrythmias
Incidence of systemic hypertension | 6 months
  Number of patients with systemic hypertension
Incidence of arterial embolism | 6 months
  Number of patients with systemic hypertension
Incidence of hemorraghe | 6 months
  Number of patients with hemorraghe
Safety mesures | 1 year
  Compare advsere events in patients with supr-ventricular arrhythmias according to the continuation or discontinuation of ibrutinib
Anticoagulants | 1 year
  Correlation between anti thrombotic strategies and cardiovascular outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Paris - Centre Université de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided